CLINICAL TRIAL: NCT01286376
Title: Randomized, Double Blind, Comparative LACTOFOS With Placebo in Constipation Patients.
Brief Title: Evaluating the Effectiveness of LACTOFOS in Constipated Patients
Acronym: COSI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Ganep Human Nutrition (Other)
Responsible Party: SKL Functional Nutrition, SKL Functional Nutrition
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COSI
Record Dates: First submitted 2011-01-20; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2010-12

CONDITIONS: Constipation
Keywords: Symbiotics; Fiber; Constipation
MeSH Terms: conditions — Constipation | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- symbiotic (Active Comparator)
  Interventions: Dietary Supplement: Symbiotic Lactofos
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Symbiotic Lactofos — Lactobacillus Paracasei Lactobacillus Rhamnosus Lactobacillus Acidophilus Bifidobacterium lactis 12g/day
  Other Names: prebiotcs; probiotcs
  Arms: symbiotic
Dietary Supplement: Maltodextrin — Maltodextrin
  Arms: placebo

SUMMARY:
Determine the effectiveness of symbiotic LACTOFOS containing FOS and probiotics against placebo in patients with a diagnosis of constipation, comparing the average number of weekly evacuations in 2 (two) groups for 30 days.

DETAILED DESCRIPTION:
A prospective, randomized, double blind, parallel group. Consist of a period of 30 days of treatment with placebo or with LACTOFOS.Will study 120 patients were female with a diagnosis of constipation according to Rome III criteria for at least 3 (three) months.

The experimental group (N = 60)will receive LACTOFOS 12g/day in two doses of 6 g. The control group (N = 60)will receive a placebo (maltodextrin) from 12g/day in two shots of 6 g.

Subsequently, the patients will be classified according to the study of AGACHAN, which determined a score based on the main complaints of patients. The symptoms that included evaluation for the total score were stool frequency, difficulty / straining, pain at defecation, feeling of incomplete evacuation, abdominal pain, time taken to initiate the evacuation, type of assistance for evacuation, failed attempts / day and duration of constipation. The intensity of each symptom varied within the range of 0 to 4, with the exception of the item type of assistance for evacuation, which ranged from 0 to 2.

Constipation is classified as mild when the total sum of values (scores) vary from 00 to 10, as moderate when the sum of the values obtained vary from 11 to 20 and severe when the final sum range from 21 to 30.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-75 years
2. A diagnosis of constipation defined by Rome III criteria
3. Ability to good communication with the investigator and agreeing to requests from the entire study
4. Patients must sign a formal consent to participate

Exclusion Criteria:

1. Constipation drug source
2. History or evidence of organic disease of the gastrointestinal tract such as tumors, inflammatory bowel disease, etc.. proven by radiological or endoscopic examination of the bowel (five years before and after onset of symptoms). If the investigator has doubts should request the necessary procedures, such as sigmoidoscopy, colonoscopy or edema bariatric to exclude organic disease
3. History of laxative use which in the opinion of the investigator is consistent with severe laxative dependence
4. Current History recent (12 months) of significant abuse of alcohol or drugs
5. History of malignancy in 5 (five) previous years (except basal cell carcinoma treated well or cervical carcinoma in situ)
6. Known history of cardiovascular control inappropriate and / or significant respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other illness which compromises the ability of patients to participate in the full study
7. Use of investigational drugs in the previous month or intentional use of such drugs during the study
8. Intention of regular use of other medications that affect intestinal motility and / or perceived
9. Lactose malabsorption is not treatable. If clinical suspicion of lactose intolerance, the procedure for proper diagnosis should be made to establish or exclude a diagnosis. If malabsorption is diagnosed, the patient should receive appropriate conditions of treatment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-03 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of stool - Chart | 30 days
  30 days taking 2 times per day. At morning and night

CONTACTS AND LOCATIONS:
Overall Officials: Dan L. Waitzberg, phd, Principal Investigator — University of Sao Paulo
Locations (1):
- Ganep Nutrição Humana, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Waitzberg DL, Logullo LC, Bittencourt AF, Torrinhas RS, Shiroma GM, Paulino NP, Teixeira-da-Silva ML. Effect of synbiotic in constipated adult women - a randomized, double-blind, placebo-controlled study of clinical response. Clin Nutr. 2013 Feb;32(1):27-33. doi: 10.1016/j.clnu.2012.08.010. Epub 2012 Aug 23. PMID 22959620